CLINICAL TRIAL: NCT04088045
Title: Exploring the Effectiveness of Combined High Frequency Intensive Autologous Platelet Rich Plasma Injection and Genicular Nerve Blocks in Treating Patients With Moderate to Severe Degrees of Knee Osteoarthritis
Brief Title: High Frequency Intensive Autologous PRP Injection and Genicular Nerve Blocks in Treating Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20100378A3
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-08

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Autologous Platelet Rich Plasma
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Patients are divided into three groups. Group 1 will receive knee IA PRP injections only. Group 2 will receive simultaneous knee IA PRP injections and PRP injections to the pes anserine complex. Group 3 will receive simultaneous knee IA PRP injections and PRP injections to the pes anserine complex, as well as to the genicular nerve blocks using 5% dextrose solution.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receiving PRP injections or PRP plus neural prolotherapy (Experimental): This experiment compares the effect of injecting PRP alone into the knee joint and pes anserinus complex with when dextrose solution is also injected to the genicular nerves.
  The injection of dextrose solution is to decrease the inflammation of the genicular nerves, hoping to further effectively alleviate the knee pain condition. Therefore, upon the conclusion of this study, we can see whether the inclusion of dextrose injection in addition to PRP treatment can really be effective in treating patients with more severe degrees of knee OA.
  Interventions: Device: Autologous platelet rich plasma and 5% dextrose solution injections.

INTERVENTIONS:
Device: Autologous platelet rich plasma and 5% dextrose solution injections. — One group of patients will receive autologous platelet rich plasma injection into the knee joint and pes anserinus complex. The other group will receive both PRP injections into the knee joint and pes anserinus complex, and prolotherapy of 5% dextrose solution to the genicular nerves.
  Dextrose solutions are injected to the genicular nerves.

SUMMARY:
Osteoarthritis (OA) of the knees is the most common degenerative disorder seen in a rehabilitation outpatient clinic. It is characterized by structural changes in the articular cartilage and the surrounding tissues. The understanding of its pathophysiology is still unclear. Knee OA patients are often troubled with knee pain and functional disturbance. Several studies have shown that the earlier the injection of autologous platelet rich plasma (PRP) to treat early stages of knee OA, the better the treatment outcome. However, there are controversies as to whether PRP injections can also be effective in treating patients with moderate to severe degrees of knee OA. Synovial fluid (SF) is in contact with the primary tissues affected by OA (cartilage and synovium). Identifying the SF biomarkers can provide us with crucial information in monitoring the PRP treatment response.

PRP is blood plasma that is rich in autologous platelets. Platelet releases growth factors and cytokines that can stimulate the healing of soft tissue structures. However, the amount of platelets in human blood is not concentrated. Purification and centrifugation procedures are needed to concentrate these platelets. The human knee cartilage is contained inside the knee joint and has scarce blood supply. When the cartilage is injured, growth factors can hardly reach this area to repair the cartilage. Therefore, many studies have suggested early usage of PRP in treating knee OA. Some studies have stated that the effect of PRP in treating knee OA is superior to that of hyaluronic acid (HA). Recent studies have recommended the application of high frequency PRP injections (ex/ intra-articular (IA) PRP injections on a weekly basis) in treating patients with more severe degrees of knee OA. Prolotherapy using hyperosmolar dextrose solution has been shown to have some positive effectiveness in treating patients with knee OA. Higher percentage, such as > 12.5% of dextrose water, may stimulate cartilage repair. Lower percentage, such as 5% dextrose water, has been documented to play an essential role in anti-inflammation, and pain reduction.

DETAILED DESCRIPTION:
Our previous study has documented that knee IA PRP injection combined with PRP injection to the pes anserine complex offered better treatment effectiveness as compared with IA PRP alone. In this two-year study, patients with moderate to severe degrees of knee OA will be recruited and divided into 3 groups. The high frequency PRP injection method will be applied (weekly PRP injections for a total of 3 weeks). Group 1 will receive knee IA PRP injections only. Group 2 will receive simultaneous knee IA PRP injections and PRP injections to the pes anserine complex. Group 3 will receive simultaneous knee IA PRP injections and PRP injections to the pes anserine complex, as well as to the genicular nerve blocks using 5% dextrose solution. We hypothesize that patients in group 3 will have better treatment outcomes. The effectiveness will be examined using proteomics, isokinetic measurements and functional scale evaluations. Upon the completion of this study, we will be able to gather adequate scientific evidences as to which injection approach and what PRP injection frequency is a better option in treating patients with moderate to severe degrees of knee OA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffered from chronic unilateral knee pain for more than 4 months and with roentgenogram degenerative findings of grades 3 and 4 on the Kellgren-Lawrence Classification of Osteoarthritis scale (meaning moderate to severe degrees of knee OA) will be recruited.
2. The volume of the SF in the supra-patellar bursa region is enough (at least 2 mm thickness in bursa fluid as measured by ultrasound) to be aspirated via ultrasound guidance.
3. Small volume of SF will be aspirated first and sent for SF analysis. SF showing evidences of crystals suggesting possible gouty arthritis and infection will not be included in this study.
4. Patient has previously received oral NSAIDs and physical modality treatments but WITHOUT any obvious improvements in knee pain and function.

The usage of musculoskeletal ultrasound to confirm that the supra-patellar bursa is in communication with the synovial cavity of the knee joint. This is to prevent the aspiration of isolated cystic lesion at the supra-patellar region.

Exclusion Criteria:

1. Total obliteration of knee joint as shown on the roentgenogram images. Patient has systemic disorders such as diabetes, rheumatoid arthritis, major axial deviation of the knee joint (varus >5°, valgus >5°), hematological diseases (coagulopathy), severe cardiovascular diseases, infections, and immune-depression.
2. Patients in therapy with anticoagulants, and taking NSAIDs within the 5 days before blood harvest
3. Patients with hemoglobin value of less than 11 g/dl, and platelet counts of less than 150,000/mm3.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Lequesne knee osteoarthritis questionnaire | About 10 minutes are required to evaluate the score of LeQuesne index.
  Lequesne knee osteoarthritis functional index includes distance, pain, and function. When added, an index score of > 7 indicates the possibility of knee osteoarthritis. The higher the score, the more severeness of knee osteoarthritis. When the index score is less than 7, the possibility of knee osteoarthritis is not high.
Two-dimensional electrophoresis (proteomics) | Two days are required to measure the protein band intensities on the gels.
  Hundreds of protein spots can be viewed on 2-dimensional electrophoresis gels. The intensity of each spot represents protein concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Carl P.C. Chen, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No